CLINICAL TRIAL: NCT04163510
Title: Family Perceptions of a Parent/Child Reading Support Program
Brief Title: Parent/Child Reading Support Program
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Because of the pandemic, this study had to be stopped and cannot be resumed.
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AAAS7425
Record Dates: First submitted 2019-11-12; First posted 2019-11-14 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Literacy
MeSH Terms: conditions — Literacy

STUDY DESIGN:
Intervention Model Description: One group of 10 sets of parents and their children will participate. The study design will use pre-intervention and post-intervention measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Reading Intervention Group (Experimental): A group of parents and their children will participate in this single arm, pre-/post-intervention study. This 10-week study will include 10 sets of parents of low-reading elementary school children, recruited from Harlem Grown Community Center. Intervention will be implemented in a 9-week period, with data collection during the first intervention week and one week post-intervention. Three large-group sessions will be held in a central location (at Harlem Grown Community Center), to build community and rapport among researchers and participants. Six individual sessions will take place in the participants' homes, to customize reading strategies and routines to each family's home setting and personal interests. The reading program will help parents identify strategies to establish literacy routines with their children, and to engage with them in enjoyable literacy activities that promote skill building while reducing negative feelings associated with reading.
  Interventions: Behavioral: Behavioral: Parent/Child Reading Program

INTERVENTIONS:
Behavioral: Behavioral: Parent/Child Reading Program — A 9-week parent/child reading program will help parents to identify strategies to establish literacy routines with their children, and to engage with them in enjoyable literacy activities that promote skill building while reducing negative feelings associated with reading. Three large-group sessions will be held in a central location, to build community and rapport among researchers and participants. Six individual sessions will take place in the participants' homes, to customize reading strategies and routines to each family's home setting and personal interests. Intervention sessions will be held once per week for 60-90 minute sessions.

SUMMARY:
Reading is a fundamental skill that is required for children's successful participation in school. Later in life, individuals who were unable to attain adequate reading levels during childhood face a cascade of deficits and social marginalization. By the end of third grade, predictions are already made about the probability of high school graduation, employability, dependence on welfare, incarceration, and decreased health outcomes. With 64% of fourth graders and 66% of eighth graders nationwide reading below grade level, illiteracy and low literacy constitute a silent epidemic that poses incredibly deleterious financial and human costs to individuals and to society. With low readers existing disproportionately in low-income communities, the children of low-income parents constitute a vulnerable sector of our society, at risk of poor literacy development and ultimately facing the above-mentioned disadvantages later in life. The purpose of this study is to empower low-income parents of elementary school children who are reading below grade level with strategies and tools to incorporate reading into their home routines; to inspire parents to approach reading with their children with an attitude of fun, positivity, and enthusiasm; to inculcate positive feelings towards reading among parents and children; and ultimately to increase the frequency of participants' home reading participation. The study will consist of a nine-week program including game playing, recipe following, neighborhood walks, trips to the library, and coaching on establishing reading resources and routines at home. Ten sets of parents will be recruited to participate in this study. Qualitative data will be extracted from field notes taken during intervention sessions and from parent interviews. It is anticipated that study results will provide information to occupational therapists to help parents better support their children's literacy development.

DETAILED DESCRIPTION:
Reading is fundamental to children's successful participation in school and a prerequisite to success in a myriad of adult occupations later in life. A student who is reading below grade level at the end of third grade is four times more likely to drop out of high school, which frequently leads to a cascade of deficits including unemployment, reduced wages, poverty, incarceration, and poor health outcomes. 64% of fourth graders and 66% of eighth graders nationwide are currently reading below grade level, with low readers existing disproportionately in low-income communities. Parental engagement in literacy activities at home with their children has decreased in recent years, thus rendering children less prepared to succeed at school. The purpose of this study is to assess a nine-week literacy support program in a low-income community, targeting the parents of elementary school children who are reading below grade level. The program intends to equip parents with strategies to incorporate literacy participation with their children into their home routines, thus increasing their children's exposure to print, reinforcing academic skills at home, and providing opportunities for positive associations with literacy. Participants will establish times in their daily schedules for reading, identify locations in their homes to organize and store reading materials, and experience a variety of pleasurable ways to engage in reading, including game playing, recipe following, neighborhood walks, and trips to the library. Ten sets of parents will be recruited to participate in this study. Qualitative data will be extracted from field notes taken during intervention sessions and from parent interviews. It is anticipated that study results will provide information to occupational therapists to help parents better support their children's literacy development.

Week 1: (Group Session at School) Meet & Greet - Food, Reading Games, Brainstorming, 60 minutes Week 2: (Group Session at School) Meet & Greet - Food, Reading Games, Introduction to Take-home Reading Kit, 60 minutes Week 3: (Home Session) Make Your Own Personal Library - Create a Bookshelf, Receive a Book & Reading Game to keep, 60 minutes

Week 4: (Home Session) Read Instructions to Create a Fun Project:

Food, Slime, Crafts Project, etc., 60 minutes

Week 5: (Home Session) Read Instructions to Create a Fun Project:

Food, Slime, Crafts Project, etc.,60 minutes Week 6: (Home Session) Library Visit & Neighborhood Word Identification Game, 90 minutes Week 7: (Home Session) Return to Library & Neighborhood Word Identification Game, 90 minutes Week 8: (Home Session) Book Making - Arts & Craft Session, 60 minutes Week 9: (Group Session at School) Wrap-up and Reinforcement - Food, Feedback & Reinforcement! 60 minutes Week 10: (Home Session) Interview and Reflection about Program, 35 minutes

ELIGIBILITY:
Inclusion Criteria:

* Participants will be parents and their children who are members of Harlem Grown Community Center.
* Elementary school children, in grades 1-3, who are having difficulty with reading skills, as perceived by their parents.

Exclusion Criteria:

* Parents who are unable to commit to a 10-week program that includes group sessions at Harlem Grown and individualized sessions in their homes will be excluded from study participation.

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Family Reading Occupations Questionnaire | week 10
  The Family Reading Occupations Questionnaire is a 14-item, 5 minute questionnaire with 4 open-ended questions and 10 Likert scale questions. The scale ranges from scores of 10 to 50 with lower scores indicating better outcomes. The questionnaire allows parents to identify the type of reading activities they engage their children with and how frequently.
Child Reading Occupations Questionnaire | week 10
  The Child Reading Occupations Questionnaire is an 8-item, 5 minute questionnaire that allows children to indicate what types of reading activities they enjoy. All questions are open-ended and provide descriptive narrative.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Gutman, PhD, Principal Investigator — Columbia University

IPD SHARING:
Plan to Share IPD: No
No plan to make individual participant data available to other researchers.